CLINICAL TRIAL: NCT01433159
Title: Comparison of HP011-101 to Standard Care in the Management of Stage I-II Pressure Ulcers in Subjects With Spinal Cord Injury
Brief Title: Comparison of HP011-101 to Standard Care for Stage I-II Pressure Ulcers in Subjects With Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011-101-09-043
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Pressure Ulcers; Spinal Cord Injury
Keywords: Pressure Ulcers; Spinal Cord Injury; Healthpoint; Xenaderm; 011-101
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HP011-101 (Experimental)
  Interventions: Drug: HP011-101 (Xenaderm Ointment)
- Various (Active Comparator): Standard Care at each site other than Xenaderm Ointment or other BCT-containing products
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: HP011-101 (Xenaderm Ointment) — The test article will be applied at approximately the thickness of a dime twice daily, or more often if removed incidental to cleansing for 14 days treatment with HP011 101.
  Arms: HP011-101
Drug: Standard Care — No restrictions are placed on the nature of this care, except that it conform to the typical practices in place during the prior 3 months and that the regimen does not include the use of a BCT ointment (ointments containing Balsam Peru, castor oil and trypsin).
  Arms: Various

SUMMARY:
The trial will compare the effects of 14 days treatment with HP011 101 versus Standard Care in subjects with Stage I or II pressure ulcers as a complication of spinal cord injury, measured as change from baseline in composite wound bed scores of the PUSH 3.0 tool.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent, or assent if less than 18 years of age.
* Age 12 years or older, of either sex, and of any race or skin type, provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* Have pressure ulcers ≤ Stage II severity, ≥ 2 cm² and ≤ 100 cm² in aggregate area (each area will be measured, including ulcer area (cm2), perimeter (cm) and greatest depth (cm) using the ARANZ Silhouette™ wound imaging and measurement device, and will remain at the treating facility for at least three weeks.
* In the opinion of the Investigator, are maintaining an adequate nutritional status and are receiving a full caloric diet, either orally or by tube.
* All female subjects must have a negative urinary pregnancy test at screening.
* Have, within 12 weeks prior to screening, clinical laboratory test results indicating:

  * Alkaline phosphatase, ALT, AST, BUN and serum creatinine levels < 3x upper limit of the Healthpoint normal range
  * HbA1C ≤ 12%
  * Hemoglobin ≥ 8 g/dL
  * Serum albumin, pre-albumin, and serum total protein measurements must be collected or obtained. These will serve as baseline covariates for analysis, but will not be used as inclusion criteria.

The most recently obtained laboratory values must be evaluated against the stated criteria. If these values are not available from a blood sample within 12 weeks of screening, blood must be drawn at screening and these laboratory values determined.

* For ulcers that will require surgical debridement, any debridement modality may be used at baseline, but the ulcer must remain a Stage I or Stage II partial thickness wound after debridement.
* Have spinal cord injuries, which are motor complete or motor incomplete injuries that are based on American Spinal Injury Association (ASIA) Impairment classifications A, B, C, and D.

Exclusion Criteria:

* Have a spinal cord injury from, epidural abscess, infection, neurodegenerative process, or malignancy.
* Have a known hypersensitivity to any of the test articles or their components.
* Have received therapy with another investigational agent within thirty (30) days of screening.
* Are pregnant or nursing.
* Have received systemic treatment with glucocorticoids for > 10 consecutive days within 1 week prior to the start of the study.
* Have received chemotherapy or radiation therapy within the past 5 years.
* Have clinical evidence of bacterial or fungal infection of the any open wound per visual/clinical assessment.
* Have a severe burn, immunodeficiency disorder, hematologic disorder, or metastatic malignancy.
* Have had documented osteomyelitis in the ulcer area within 6 months prior to screening.
* Have end-stage renal disease, are receiving treatment for cancer (except for non-melanoma skin cancer within the past five years), or untreated peripheral vascular disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (5):
- United States (5):
  - VA Medical Center, Long Beach, Long Beach, California
  - Santa Clara Valley Medical Center, San Jose, California
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - Carolinas Research, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects >/= 12 yrs of age with Stage I or II pressure ulcers between 1 and 100 cm2 (inclusive) in total aggregate area and maintaining an adequate nutritional status and were receiving a full caloric diet, either orally or by tube
Groups:
- HP011-101: Xenaderm Ointment
- Various Standard Care: Standard Care at each site other than Xenaderm Ointment or other BCT2-containing products
Period: Overall Study
Arm/Group | HP011-101 | Various Standard Care
Started | 9 | 10
Completed | 7 | 9
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HP011-101 | Various Standard Care | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (20.7) | 58.6 (18.4) | 57.4 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Composite PUSH (Pressure Ulcer Scale for Healing) Score
Description: Change from baseline in composite wound bed scores measured as the PUSH total score on Day 15. The PUSH Tool v.3.0, which monitors the three critical parameters that are the most indicative of healing, was used in this study. Scales for the three measurements were: Area = 0 (healthy skin) to 10 (>24 cm x cm); Exudate = 0 (non) to 3 (heavy); Tissue type = 0 (epithelial tissue) to 4 (necrotic tissue). All values were summed and final values are the cumulative scores.
  Cumulative Scores = 0 (Best possible outcome: healthy skin/epithelial tissue with no exudate) to 17 (Worst possible outcome: wound >24 cm x cm, containing necrotic tissue, with heavy exudate)
Time Frame: baseline, 14 Days
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Groups:
- Various Standard Care: Standard Care at each site other than Xenaderm Ointment or other BCT-containing products
Arm/Group | HP011-101 | Various Standard Care
Number analyzed (Participants) | 7 | 9
scores on a scale | -3.20 (2.00) | -3.47 (3.73)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | HP011-101 | Various Standard Care
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP011-101 (N=9) | Various Standard Care (N=10)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject developed a second pressure ulcer near target ulcer and discontinued from the study in error by Investigator. Discontinuation resulted in protocol deviation as subject could have remained in the study and was not required to be discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less